CLINICAL TRIAL: NCT00277732
Title: Pharmaceutical Care for Diabetes Type 2 Patients: a Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005/340
Record Dates: First submitted 2006-01-13; First posted 2006-01-16 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Pharmaceutical care at baseline and follow-up visits over 6 months

SUMMARY:
The objective of this study is to evaluate the therapeutic effectiveness and cost-effectivity of pharmaceutical care for diabetes type 2 patients. Patients will be randomly allocated to the control group ( = no input from pharmacist) or intervention group ( = with pharmaceutical care at baseline and follow-up visits over 6 months).

ELIGIBILITY:
Inclusion Criteria:

* 45-75 years
* Body Mass Index >= 25
* Diabetes treatment for at least 12 months
* Regular visitors of the participating community pharmacy

Exclusion Criteria:

* Patients taking only insulin (no oral antidiabetic drugs)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2006-01; Study Completion 2006-11

PRIMARY OUTCOMES:
The difference between the study groups in the change of blood glucose and HbA1c | baseline and after 6 months

SECONDARY OUTCOMES:
Knowledge about diabetes and treatment | after 6 months
Therapy adherence
Body Mass Index | after 6 months
Periods of severe hypoglycemia
GP visits, emergency room visits and hospitalisations
Work days lost
Frequency of eye and foot examination

CONTACTS AND LOCATIONS:
Overall Officials: Mimi Giri, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Ghent — http://www.ugent.be